# **Study Plan of**

PROSPECTIVE, RANDOMIZED, CONTROLLED, DOUBLE-BLIND, MULTI-CENTRIC, INTERNATIONAL STUDY ON THE EFFICACY AND SAFETY OF AN EARLY TARGET CONTROLLED PLASMA VOLUME REPLACEMENT THERAPY WITH A BALANCED GELATIN SOLUTION VS A BALANCED ELECTROLYTE SOLUTION IN PATIENTS WITH SEVERE SEPSIS / SEPTIC SHOCK

**GENIUS (GELATIN IN ICU AND SEPSIS)** 

STUDY IDENTIFICATION NO.: HC-G-H-1209

# NCT02715466

Date of final applicable study plan: 16.06.2020

**Marketing Authorization Holder:** 

B. Braun Melsungen AG Germany

Organized and Financed by:

B. Braun Melsungen AG Division Hospital Care Carl-Braun-Str. 1 34212 Melsungen Germany

# STUDY OVERVIEW

| Title of Study | PROSPECTIVE, RANDOMIZED, CONTROLLED, DOUBLE-BLIND, MULTI-CENTRIC, INTERNATIONAL STUDY ON THE EFFICACY AND SAFETY OF AN EARLY TARGET CONTROLLED PLASMA VOLUME REPLACEMENT THERAPY WITH A BALANCED GELATIN SOLUTION VS A BALANCED ELECTROLYTE SOLUTION IN PATIENTS WITH SEVERE SEPSIS / SEPTIC SHOCK |
|---|---|
| Acronym | GENIUS (GELATIN IN ICU AND SEPSIS) |
| Investigational Products (IPs) | <ul> <li>Investigational test product (gelatin group): Gelaspan (plasma adapted gelatin solution for infusion)</li> <li>To be administered in combination with background medication (i.e. open-label Sterofundin ISO; a plasma adapted electrolyte solution) in a ratio of 1:1 (gelatin:electrolyte)</li> </ul> |
| | <ul> <li>Investigational reference product (crystalloid group): Sterofundin ISO (plasma adapted electrolyte solution)</li> <li>To be administered in combination with background medication (i.e. open-label Sterofundin ISO; a plasma adapted electrolyte solution) in a ratio of 1:1</li> </ul> |
| Background Medication | Open-label Sterofundin ISO (plasma adapted electrolyte solution) |
| Phase | IV |
| Study Design | Prospective, controlled, randomized, double-blind, international, multi-centric study with two parallel groups |
| Number of Sites & Countries | Multi-centric, international (Participating countries: Austria, Czech Republic, France, Germany, Spain) Up to 15 sites |
| Sample Size | 2 x 304 patients (in total 608 patients) |
| | Sample size re-calculation after 2 x 200 (in total 400) patients. |
| Indication | Hypovolaemia in Severe Sepsis / Septic Shock |
| Primary Objective | Investigate the efficacy of early goal directed fluid management of a combination of a gelatin and crystalloid regime in comparison to a pure crystalloid regime in achieving haemodynamic stability (HDS) in patients with severe sepsis / septic shock. |
| Primary Variable | Time until first / initial HDS is achieved (in minutes). |
| | Time measurement will start with first administration of IPs and will be continued until first HDS is achieved. |
| Secondary Objectives | Investigation of safety and efficacy parameters of the applied fluid regimes. |
| Secondary Variables | <ul> <li>Safety</li> <li>Renal function</li> <li>Serum creatinine (SCr)</li> <li>Serum blood urea nitrogen (BUN)</li> <li>Estimated glomerular filtration rate (eGFR)</li> <li>Need and indication of renal replacement therapy (RRT)</li> </ul> |

- Urine output
- Kidney Disease Improving Global Outcome (KDIGO) score

#### Coagulation

- Prothrombin time (PT)
- Activated partial thromboplastin time (aPTT)
- International norm ratio (INR)

Site specific measurements (Innsbruck):

- Fibrinogen
- Antithrombin (AT)
- Platelets absolute

#### Hepatic function

Bilirubin

#### Adverse Events

• (Serious) adverse events ((S)AEs) / reactions ((S)ARs)

#### Other

- Number of red blood cell (RBC) units
- Number of fresh frozen plasma (FFP) units
- Number of other blood products
- Vasopressor therapy
- Inotropic therapy

# Efficacy

Fluid administration according to the volume algorithm

- Volume needed to achieve first / initial HDS
- Total volume until 48 h after randomization
- Administered bottles

Additional administered crystalloid solutions for further volume treatment

Drug and volume

#### Fluid balance

- Fluid intake
- Fluid output
- Fluid balance

# Haemodynamics

- Volume responsiveness upon passive leg raising (PLR) or exogenous fluid challenge
- Haemodynamic readings as required by the volume algorithm and haemodynamics from 48 h after randomization until ICU discharge or day 28, whatever occurs first

Tissue oxygenation and acid base balance

Arterial blood gas analyses (BGA)

- Serum electrolytes
- Base excess (BE)
- Lactate / lactate decrease
- Central venous BGA
- Arterial oxygen content
- Oxygen delivery

#### • Outcome

- Length of stay (LOS) in the intensive care unit (ICU)
- Hospital LOS
- Days on RRT
- Number of infection free days
- Number of antibiotic free days
- Number of ventilator free days
- Number of vasopressor free days

#### • Follow-up

- Last available SCr (day 28)
- Colloid therapy (day 28)
- Mortality & cause of death (if applicable) (day 28 & day 90)
- Health-related quality of life (HRQoL) (day 90)
- New RRT / kidney disease (day 90)

#### • Other variables

# Demographic data

- Age
- Gender
- Height
- Weight
- Race
- Type of patient (e.g. trauma patient, surgical patient)

#### Anamnesis

- APACHE II & SOFA score
- Temperature
- Fluid input in the 24 h prior to randomization
- Origin of sepsis
- Procalcitonin (optional)
- Causative organism of infection
- Medical history

#### Concomitant medication

- Antibiotic therapy
- Nephrotoxic therapy
- Contrast agents
- Anticoagulation therapy

#### Study termination

# Patient Inclusion / Exclusion Criteria

#### Inclusion criteria:

- Male or female patients ≥ 18 years of age
- Women of child bearing potential must test negative on standard pregnancy test (urine or serum)
- Patients with body weight  $\leq 140 \text{ kg}$
- Patients diagnosed severe sepsis / septic shock (refer to section Fehler!
   Verweisquelle konnte nicht gefunden werden. for definitions) at
   admission on ICU who can be enrolled within 90 min after admission OR
   patients diagnosed severe sepsis / septic shock during ICU stay who can
   be enrolled within 90 min after diagnosis
- Patients where antibiotic therapy has already been started (prior to randomization)
- Patients who are fluid responsive. Fluid responsiveness is defined as increase of > 10% in mean arterial pressure (MAP) after PLR or fluid challenge (max. 250 ml crystalloid solution)
- Signed informed consent by patient, legal representative or authorized person or deferred consent

#### Exclusion criteria:

- Administration of HES, dextrane solutions or > 500 ml of Gelatin solutions within the 24 h prior to randomization
- Death expected within the next 48 h (moribund patients as defined by ASA ≥ class V)
- Patients with confirmed acute SARS-CoV-2 (COVID-19) infection (as available from routine medical records/ patient chart)
- Patients for whom the need of pressure infusions are expected
- Requirement for renal support (either continuous or discontinuous techniques, including intermittent haemodialysis, haemofiltration and haemodiafiltration)
- Patients receiving therapeutic heparin medication due to chronic coagulation disease / anticoagulation medication (i.e. partial thromboplastin time > 60 sec)
- Acutely burned patients (refer to section )
- Renal failure with oliguria or anuria
- Severe general oedema
- Severe congestive cardiac failure
- Hypersensitivity to the active substance or ingredients of the IPs
- Hypersensitivity to galactose-α-1,3-galactose (alpha-Gal) or known allergy to red meat (mammal meat) and offal
- Hypervolaemia / hyperhydration
- Hyperkalaemia
- Hypercalcaemia
- Metabolic alkalosis

| | Simultaneous participation in another interventional medical devices studies) | clinical trial (drugs o |
|---|---|---|
| Investigational Test<br>Product | Gelaspan: Plasma adapted gelatin solution for infusion Composition (1000 ml solution contain): | |
| | Succinylated gelatin (= modified fluid gelatin) | 40.0 g |
| | Sodium chloride | 5.55 g |
| | Sodium acetate trihydrate | 3.27 g |
| | Potassium chloride | |
| | | 0.30 g |
| | Calcium chloride dihydrate | 0.15 g |
| | Magnesium chloride hexahydrate | 0.20 g |
| | Excipients for pH-adjustment: | |
| | Sodium hydroxide 40% | 0 - 0.133 g |
| | Hydrochloric acid 20% | 0 - 0.182 g |
| | Electrolyte concentrations | |
| | Sodium | 151 mmol/l |
| | Chloride | 103 mmol/l |
| | Potassium | 4 mmol/l |
| | Calcium | 1 mmol/l |
| | Magnesium | 1 mmol/l |
| | Bicarbonate as Acetate | 24 mmol/l |
| | Molecular weight, weight average: | 30 000 Dalton |
| | | 23 200 Dalton |
| | Molecular weight, number average: Theoretical osmolarity: | 284 mOsm/l |
| Investigational Reference | Sterofundin ISO: Plasma adapted electrolyte solution fo | |
| Product | Composition (1000 ml solution contain): | |
| | Sodium chloride | 6.80 g |
| | Potassium chloride | $0.30 \mathrm{g}$ |
| | Calcium chloride dihydrate | $0.37~\mathrm{g}$ |
| | Magnesium chloride hexahydrate | 0.20 g |
| | Sodium acetate trihydrate | 3.27 g |
| | Malic acid | 0.67 g |
| | Electrolete consentration | C |
| | Electrolyte concentration | 1.45.0 1/1 |
| | Sodium | 145.0 mmol/l |
| | Potassium | 4.0 mmol/l |
| | Calcium | 2.5 mmol/l |
| | Magnesium | 1.0 mmol/l |
| | Chloride | 127.0 mmol/l |
| | Acetate | 24.0 mmol/l |
| | Malic acid | 5.0 mmol/l |
| | pH: | 5.1 - 5.9 |
| | Theoretical osmolarity: | 309 mOsmol/l |
| Fluid Administration | Method of Administration The administration of IPs and background medication is performed intravenously. | |
| | Dosage | |

Dosing of IPs is individualized to the patient's volume needs. Blinded IP volume applied should not exceed 30 ml/kg/day.

In addition background medication is applied alternating with IPs in a ratio of 1:1.

Fluids are administered according to the volume algorithm as long as the patient is fluid responsive. Fluid responsiveness is defined as an increase of 10% of MAP and / or stroke volume index (SVI) after endogenous or exogenous fluid challenge. An endogenous fluid challenge is achieved by means of PLR. An exogenous fluid challenge is achieved by infusing 500 ml of fluid in 15 min.

Refer to protocol section  for details on the fluid management strategy.

#### **Duration of Treatment**

Treatment with IPs starts directly with randomization and discontinues with the achievement of HDS, achievement of maximum daily dose (30 ml/kg) or 48 h after randomization, whatever occurs first.

#### Visit Schedule

### Prior randomization - 90 min window:

- Verification of in- / exclusion criteria
- RBC and antibiotic therapy prior randomization
- Demographic data including pregnancy test in women of childbearing potential
- Anamnesis & medical history

#### At randomization

• Blood samples for laboratory evaluations (renal function, coagulation, hepatic function, lactate, scores) - immediately before first IP administration

#### Randomisation until 48 h thereafter:

- Set of catheters (e.g. arterial line, central-venous line)
- Set of urinary catheter
- Assessment of HDS and primary endpoint 'time to first / initial HDS' (lactate, urine production, ScvO<sub>2</sub>)
- SCr (every 6 h until 48 h after randomization)
- Urine output (every 6 h until 48 h after randomization)
- Blood samples for laboratory evaluations (renal function, coagulation, hepatic function)
- Vasopressor therapy
- Inotropic therapy
- Fluid administration (i.e. IP and background medication acc. to volume algorithm)
- Administered crystalloids for further volume treatment
- Fluid intake & fluid output
- Fluid responsiveness upon PLR or exogenous fluid challenges as required by the volume algorithm
- Haemodynamic readings as required by the volume algorithm

- Tissue oxygenation and acid base balance (BGA within the first 6 h every 2 h, then every 12 h until 48 h after randomization)
- (Serious) adverse events / reactions
- Applied blood products
- Concomitant medications
- SOFA score, temperature
- Fulfilment of ICU discharge criteria
- RRT including indication
- Invasive mechanical ventilation

# 48 h after randomization until ICU discharge or day 28 (whatever occurs first):

- Blood samples for laboratory evaluations (renal function, coagulation, hepatic function)
- Severe sepsis / septic shock (second, third,... hit)
- Vasopressor therapy
- Inotropic therapy
- Administered crystalloids for further volume treatment
- Fluid intake & fluid output
- Urine output
- Haemodynamic readings (minimum and maximum daily)
- Tissue oxygenation and acid base balance
- (Serious) adverse events / reactions
- Applied blood products
- Concomitant medications
- SOFA score, temperature
- Fulfilment of ICU discharge criteria
- RRT including indication
- Invasive mechanical ventilation
- Several outcome parameters (hospital LOS, ICU LOS, number of ventilator free days, number of infection free days, number of antibiotic free days, number of vasopressor free days, days on RRT)
- Study termination

# Day 28:

- Last available SCr documented from ICU discharge until hospital discharge or day 28, whatever occurs first
- Colloid therapy from ICU discharge until hospital discharge or day 28, whatever occurs first
- Mortality & cause of death if applicable

#### Day 90:

- Mortality & cause of death if applicable
- New RRT / kidney disease

| | HRQoL questionnaire & appendix (if applicable) |
|---|---|
| Duration of Study per<br>Patient | Start of study: With randomization Treatment period (administration of fluids according to the volume algorithm): • Start of administration: With randomization |
| | Duration of administration: |
| | <ul> <li>Treatment with fluids according to the volume algorithm<br/>discontinues with the achievement of HDS or 48 h after<br/>randomization, whatever occurs first</li> </ul> |
| | <ul> <li>Treatment with additional crystalloid solutions for further volume<br/>treatment only starts after achievement of HDS, achievement of<br/>max. daily dose or 48 h after randomization until ICU discharge or<br/>day 28, whatever occurs first</li> </ul> |
| | End of study: ICU discharge or day 28, whatever occurs first Follow ups: day 28 & day 90 |
| Study Schedule | Planned start: Q1 / 2016 |
| | Planned recruitment time: 5.5 years |
| | Planned last patient out: Q4 / 2021 |
| Statistical Methods | Sample size will be based on assumption of difference between the gelatin and the crystalloid group. |
| Randomization / Blinding | Randomized with the following strata: • Site |
| | RBCs pre-treatment within 24 h prior to randomization |
| | Double-blinded |
| Data Safety Monitoring<br>Board (DSMB) | A DSMB is appointed. |